CLINICAL TRIAL: NCT02421458
Title: Dutch Randomized Multicenter Trial COmparing twO PalliativE RAdiaTION Schemes for Incurable Head and Neck Cancer (COOPERATION)
Brief Title: Comparing Two Palliative Schemes of Radiotherapy for Head and Neck Cancer
Acronym: COOPERATION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting rate was to low
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15CRH
Record Dates: First submitted 2015-02-12; First posted 2015-04-20 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1: 6 fractions of radiation (Active Comparator): radiation in a 6 fractions scheme and a daily dose of 6 Gy
  Interventions: Radiation: 6 x 6 Gy
- arm 2: 16 fractrions of radiation (Active Comparator): radiation in a 16 fractions scheme and a daily dose of 3.125 Gy
  Interventions: Radiation: 16 x 3.125 Gy

INTERVENTIONS:
Radiation: 6 x 6 Gy — radiation in 6 fraction of 6 Gy, twice a week during 3 weeks
  Arms: arm 1: 6 fractions of radiation
Radiation: 16 x 3.125 Gy — radiation in 16 fraction of 3.125 Gy, 4 times a week during 4 weeks
  Arms: arm 2: 16 fractrions of radiation

SUMMARY:
RCT to compare two radiation schemes for palliative HeadNeck cancer

DETAILED DESCRIPTION:
A substantial proportion of patients with head and neck (HNC) are not suitable for curative treatment with surgery and/or (chemo)radiotherapy (CRT) because of very advanced stage, significant comorbidities, bad general condition, distant metastasis, or a combination of these factors. Although radiotherapy (RT) is a commonly used option to achieve durable disease control and to alleviate troublesome symptoms, the data about the optimal radiation scheme and the impact of these schedules on quality of life (QoL) of these vulnerable patients is extremely scarce.

Although different radiation schemes are used worldwide (in the Netherlands, at least 15 different radiation schedules are used), it is currently not possible to identify the best RT scheme, based only on retrospective studies because of the major differences between these studies with regard to patient's demographics, radiation schedules given, the radiation technique used etc. Furthermore, no any information is available on the impact of these schemes on treatment-related toxicity and QoL.

This illustrates the urgent need for a multicenter randomized controlled trial (RCT) to identify the most optimal schemes of RT for this group of patients. Therefore, the investigators intend to initiate a prospective RCT comparing the survival, loco-regional control, toxicity, and QoL of two commonly used schemes. This study will be the first of his kind for palliative patients with HNC and will compare a short-course (6 fractions) with a long-course of radiotherapy (16 fractions). Because most of patients with incurable HNC have a poor performance status and major comorbidity and prefer limited number of visits to the hospital, it is quite reasonable to investigate whether a short scheme of radiotherapy with limited number of visits to the clinic as good as a relatively long-course of radiotherapy in terms of outcome, toxicity and QoL. This delicate balance between outcomes, possible toxicity and patient's comfort would justify the initiation of such randomized trial. The results of this study will in the nearby future enable us to indicate the radiation scheme best suits which patient category

ELIGIBILITY:
Inclusion Criteria:

• Newly diagnosed patients with primary non-metastatic carcinoma located in the oral cavity, oropharynx, larynx (except T1 glottic), hypopharynx, nasopharynx, paranasal sinuses and salivary gland and carcinoma of unknown primary in the head and neck region who are not suitable for radical treatment with surgery or (chemo) and, therefore, planned for treatment with radiotherapy in palliative setting.

OR

* Newly diagnosed patients with primary head and neck carcinoma with limited metastatic disease in a good general condition and few comorbidities (ACE-25 <3) with life expectancy of at least 6 months are also eligible.
* No chemotherapy or surgery is allowed before inclusion.
* Age ≥ 18 years
* WHO performance status 0-2
* Signed written informed consent

Exclusion Criteria:

* Patients with previously radiation treatment in the head and neck region, for any reason.

  * Chemotherapy or surgery for head and neck tumor before inclusion and no other concomitant anti-cancer therapy is allowed during study treatment.
* Patients with head and neck malignancies arising from skin, nose, thyroid gland or esophagus.
* Patients with advanced stage sarcoma or lymphoma of the head and neck region.
* Expected life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
time to loco-regional progression | 4 months
  caculated from date of response until the date of clinical deteriotion; accoriding to RECIST
impact of both radiation schemes on QoL | 2 years
  this will be measured by the EORTC questionnaires C30 and HN35; analysis will be performed by a random effects regression model

SECONDARY OUTCOMES:
overall survival rates | 4 months
  RECIST
loco-regional control rates | 3 months
  caculated from date of response until the date of clinical deteriotion; according to RECIST
overall response rates | 2 year
  caculated from date of response until the date of clinical deteriotion; accoriding to RECIST
compliance to the study treatments as assessed by completed treatment and follow-up visits | 4 months
  number of treatment fractions and follow-up visits
the incidence of grade ≥ 2 acute and late toxicity | 2 years
  scoring of AE according tot CTC 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Abrahim Al-Mamgani, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (11):
- Netherlands (11):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Radiotherapiegroep, lokatie Arnhem, Arnhem
  - University Medical Center Groningen, Groningen
  - Maastro Clinic, Maastricht
  - Radboud umc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - Instituut Verbeeten, Tilburg

REFERENCES:
- [Derived] Al-Mamgani A, Kessels R, Verhoef CG, Navran A, Hamming-Vrieze O, Kaanders JHAM, Steenbakkers RJHM, Tans L, Hoebers F, Ong F, van Werkhoven E, Langendijk JA. Randomized controlled trial to identify the optimal radiotherapy scheme for palliative treatment of incurable head and neck squamous cell carcinoma. Radiother Oncol. 2020 Aug;149:181-188. doi: 10.1016/j.radonc.2020.05.020. Epub 2020 May 14. PMID 32417345